CLINICAL TRIAL: NCT01093872
Title: Repetitive Transcranial Magnetic Stimulation for Tinnitus Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #2008/061/A
Record Dates: First submitted 2010-03-24; First posted 2010-03-26 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-08

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — Upon recruitment, all patients will undergo a 1 week treatment consisting of 5 rTMS sessions
  Repetitive TMS consists of 1000 stimulations/ day at 1 Hz and 110% of the motor threshold, for five consecutive days over the left AC.

SUMMARY:
In this study, we perform an open-label rTMS over the left AC on patients with tinnitus. Outcome measures will be evaluated statistically. The results will be instrumental in deciding the efficacy of this technique in a local patient group.

DETAILED DESCRIPTION:
Tinnitus is a subjective auditory perception of sounds or noise not triggered by external auditory stimuli, affecting millions of people worldwide. To date, pharmacological and physical/ behavioural treatments in severe cases are generally unsatisfactory. Functional brain imaging changes associated with tinnitus include hyperactivity of discrete temporoparietal regions, including both the primary auditory cortex (AC) and the secondary, or associative cortex. High-frequency rTMS (10 Hz or more) applied on the scalp overlying the hyperactive left AC produced an intense tinnitus attenuation.

Repetitive TMS consists of 1000 stimulations/ day at 1 Hz and 110% of the motor threshold, for five consecutive days over the left AC. A high number of stimuli/day were applied because of the previously suggested dose dependency of tinnitus alleviation by rTMS. Furthermore, the use of such relatively high intensity assured the stimulation of most of the target region, even in the case of mismatch between the scalp position and the underlying anatomy, which can be expected using the International EEG system as anatomical reference for TMS stimulation.

Upon recruitment, all patients will undergo a 1 week treatment consisting of 5 rTMS sessions. Tinnitus rating will be performed weekly.

Tinnitus is rated by a 0-100 Visual Analogue Scale (VAS), where 0 is wellness and 100 the worst possible tinnitus related discomfort. In addition, our validated Tinnitus Inventory scoring will be administered. Audiometry and otoscopy will be performed at enrolment and at the end of the study. Tinnitus, and acoustic evaluations are then collected by experimenters blind to the type of rTMS applied.

Standard statistical methods (SPSS for Windows) will be used to perform comparisons.

ELIGIBILITY:
Inclusion Criteria:

* All patients with tinnitus

Exclusion Criteria:

* Patients with contraindications to TMS: pacemaker, intracranial surgery, implants and seizures

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-08; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Tinnitus Inventory Handicap scoring & Visual Analogue Scale (VAS) | Baseline, 1,2,3 & 4weeks after treatment
  THI and VAS is measure before the treatment and weekly for 4 weeks after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: YL Lo, MD, Principal Investigator — National Neuroscience Institute, Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Outram Road, Singapore